CLINICAL TRIAL: NCT02660060
Title: Bioequivalence Study of 0.25 mg Pramipexole Tablets Produced by PT Dexa Medica for PT Ferron Par Pharmaceuticals in Comparison With the Comparator Product (Sifrol® 0.25 mg Tablet, Boehringer Ingelheim Pharma GmbH & Co. KG, Germany for Boehringer Ingelheim International, GmbH, Germany)
Brief Title: Bioequivalence Study of Two Formulations of Pramipexole Tablets 0.25 mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PR.193/EQL/2010
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Pramipexole; Bioequivalence; Pharmacokinetics
MeSH Terms: interventions — Pramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pramipexole Dexa Medica (Experimental): Each tablet contains 0.25 mg pramipexole dihydrochloride monohydrate. An oral single dose of the tablet was administered at the first day of each treatment period.
  Interventions: Drug: Pramipexole Dexa Medica
- Pramipexole Boehringer Ingelheim Pharma (Active Comparator): Each tablet contains 0.25 mg pramipexole dihydrochloride monohydrate. An oral single dose of the tablet was administered at the first day of each treatment period.
  Interventions: Drug: Pramipexole Boehringer Ingelheim Pharma

INTERVENTIONS:
Drug: Pramipexole Dexa Medica — Pramipexole 0.25 tablets produced by PT Dexa Medica for PT Ferron Par Pharmaceuticals as the test drug.
  Arms: Pramipexole Dexa Medica
Drug: Pramipexole Boehringer Ingelheim Pharma — Pramipexole 0.25 tablets produced by Boehringer Ingelheim Pharma GmbH & Co.KG for Boehringer Ingelheim International GmbH as the reference drug.
  Other Names: Sifrol®
  Arms: Pramipexole Boehringer Ingelheim Pharma

SUMMARY:
The present study was conducted to find out whether the bioavailability of 0.25 mg pramipexole tablets produced by PT Dexa Medica for PT Ferron Par Pharmaceuticals was equivalent to the reference drug (Sifrol® tablet 0.25 mg, Boehringer Ingelheim Pharma GmbH & Co. KG, Germany for Boehringer Ingelheim International GmbH, Germany).

DETAILED DESCRIPTION:
This was a randomized, open label, two-period, two-sequence, crossover study under fasting condition. The participating subjects were required to have an overnight fast and in the next morning were given orally one tablet of the test drug (Pramipexole 0.25 mg produced by PT Dexa Medica for PT Ferron Par Pharmaceuticals) or one tablet of the reference drug (Sifrol® 0.25 mg, Boehringer Ingelheim Pharma GmbH & Co. KG, Germany for Boehringer Ingelheim International GmbH, Germany).

Blood samples were drawn immediately before taking the drug (control), at 20, 40 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours after drug administration. Seven days after the first drug administration (washout period), the procedure was repeated using the alternate drug. The plasma concentrations of pramipexole were determined by validated ultra performance liquid chromatography with mass spectrometry detector (UPLC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* Preferably non-smokers or smoke less than 10 cigarettes per day
* Body mass index within 18 to 25 kg/m2
* Normal vital signs (after 10 minutes rest): systolic blood pressure 100 - 120 mmHg, diastolic blood pressure 60 - 80 mmHg, pulse rate 60 - 90 bpm

Exclusion Criteria:

* Personal / family history of allergy or hypersensitivity or contraindication to pramipexole or allied drugs
* Pregnant or lactating women
* Any major illness in the past 90 days or clinically significant ongoing chronic medical illness
* Any clinically significant abnormal values of liver function test (ALT, alkaline phosphatase, total bilirubin >= 1.5 upper limit normal), renal function test (serum creatinine > 1.4 mg/dL), etc
* Positive Hepatitis B surface antigen (HbsAg), anti-HCV, or anti-HIV
* Clinically significant hematology abnormalities
* Clinically significant ECG abnormalities
* Any surgical or medical condition (present or history) which might significantly alter the pharmacokinetics of the study drug
* History of anaphylaxis or angioedema
* History of drug or alcohol abuse within 12 months prior to screening
* Participation in any clinical trial within the past 90 days
* History of any bleeding or coagulative disorders
* History of difficulty with donating blood or difficulty in accessibility of veins in left or right arm
* A donation or loss of 300 mL (or more) of blood within 3 months before the study's first dosing day
* Intake of any prescription, non-prescription drug, food supplement or herbal medicine within 14 days of the study's first dosing day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
AUCt | 48 hours
  Area under plasma concentration time curve from time zero to the last observed quantifiable concentration was determined from plasma concentrations of pramipexole from the test drug and reference drug.
AUCinf | 48 hours
  Area under plasma concentration time curve from time zero to infinity was determined from plasma concentrations of pramipexole from the test drug and reference drug.
Cmax | 48 hours
  The peak plasma concentration of the drug was determined from plasma concentrations of pramipexole from the test drug and reference drug.

SECONDARY OUTCOMES:
Tmax | 48 hours
  The time needed to achieve the peak plasma concentration was determined from plasma concentrations of pramipexole from the test drug and reference drug.
T1/2 | 48 hours
  The elimination half life was determined from plasma concentrations of pramipexole from the test drug and reference drug.

CONTACTS AND LOCATIONS:
Overall Officials: Ratih SI Putri, MD, Principal Investigator — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No